CLINICAL TRIAL: NCT02602002
Title: Experimental Medicine Study to Validate Pharmacodynamic Pain Assessments in Healthy Volunteers in a Randomised, Double Blind, Placebo Controlled, 2 Way Cross-over Design With an Opioid Analgesic (Remifentanil)
Brief Title: Experimental Medicine Study to Validate Pharmacodynamic Pain Assessments in Healthy Volunteers With an Opioid Analgesic (Remifentanil)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 111000
Record Dates: First submitted 2012-04-19; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Pain
Keywords: Remifentanil, Pharmacodynamic Pain assessments, Intravenous, South Korea
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Remifentanil 0.1 ug/kg/min to 0.10 ug/kg/min
  Interventions: Drug: Remifentanil
- Placebo (Placebo Comparator): Saline (0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remifentanil — IV
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This was a single centre, randomised, double blind, placebo controlled, two-way cross-over design study to assess the feasibility of pain PD tests and to determine the variability and effects of a known analgesic drug (the opioid remifentanil) in South Korean healthy volunteers.

DETAILED DESCRIPTION:
Pain is an area of large unmet medical need and a priority disease area for GlaxoSmithKline. Selection of new candidates for pain involves tests in animal models; however, their predictive value may be limited. High risks are carried forward into Phase II Proof of Concept (PoC) studies that require large financial and time commitments.

Assessment of pain in Phase I studies can serve as a useful indicator of pharmacodynamic activity of potential analgesic treatments to reduce development risks, help make decisions about further compound progression, dose selection and design of clinical studies in pain patients. GlaxoSmithKline's Pain & Neurophysiology group at Clinical Unit Cambridge (CUC) has developed a number of human pain models specifically tailored for GSK's portfolio and began their implementation into clinical development. Some of these models have already been used successfully to detect PD activity in Phase I [Chizh, 2007] Currently, for most candidates selected by the neurology Centre for Excellence in Drug Discovery (CEDD, there are plans to utilise human pain models as part of clinical development, including FTIH studies. Because of the limited in-house capacities, there is an ongoing effort to identify a suitable external group(s) to which some of the methodologies in pain models and PD assessments could be transferred. Involving such external groups could also help access new patient groups, such that Phase I and Phase II experimental assessments could be facilitated to provide early indication of efficacy before large scale multi-centre trials are initiated.

South Korea has been identified as a country within the Asia-Pacific region to which GlaxoSmithKline would like to collaborate more closely in terms of early phase clinical trials, particularly First Time in Human studies. A satisfactory validation study will enable us to use these methodologies in future pain studies in order to link early efficacy assessments (Phase I) with future patient studies (Phase II) within South Korea.

One group that has been identified is the Clinical Trials Center of Seoul National University Hospital. This site is being considered to perform a number of clinical studies of potential new treatments for pain.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy adult male, aged 20-45 years inclusive.
* Body weight >50 Kg and BMI within the range 18.5-29.9 Kg/m2 inclusive
* Healthy as judged by a responsible physician. No clinically significant abnormality identified on the medical or laboratory evaluation. A subject with a clinically significant abnormality or laboratory parameters outside the reference range for the relevant age group may be included only if the Investigator and Medical Monitor consider that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* A normal 12-lead ECG recording at the pre-study medical.
* Signed and dated written and informed consent must be obtained for all subjects prior to admission to the study.
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* The subject has a positive pre-study urine screen for drugs of abuse or positive alcohol test.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. 1 unit is equivalent to a half-pint (220 mL) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine.
* Use of prescription drugs as well as vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless it is the opinion of the Investigator and Medical Monitor that the medication will not interfere with the study procedures or compromise subject safety.
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* Has a systolic blood pressure which is outside the range of 90 to 140 mmHg, diastolic blood pressure is outside the range of 50 to 90 mmHg or heart rate is outside the range 40 to 90 bpm.
* Has a QTcB >450 msec.
* Has a significant medical history of dizziness, blackouts, fainting or vaso-vagal attacks.
* Has received over-the-counter (OTC) medicine within 48h before the first dosing day. Subjects who have taken OTC medication may still be entered into the study, if, in the opinion of the Principal/Co-Investigator, the medication received will not interfere with the study procedures or compromise safety.
* Has a history or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the distribution, metabolism or excretion of drugs.
* The subject has received an investigational drug or participated in any other research trial within 84 days for new chemical entities and marketed drugs or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To measure the Heat Pain Threshold of a marketed opioid analgesic versus placebo on quantitative experimental pharmacodynamic pain markers. | pre-dose to 67 mins
  Heat pain threshold

SECONDARY OUTCOMES:
To measure the Mechanical Pain Threshold of a marketed opioid analgesic versus placebo. on quantitative experimental pharmacodynamic pain markers. | Change from Baseline (pre-dose) in mechanical pain thresholds measurements at 46 minutes
  Mechanical pain threshold measurements (von Frey filaments) reported by treatment group and dose levels.
To measure the Pressure Pain Threshold of a marketed opioid analgesic versus placebo on quantitative pharmacodynamic experimental pain markers. | Change from Baseline (pre-dose) in mechanical pain thresholds measurements at 46mins
  Mechanical pain threshold measurements (von Frey filaments) reported by treatment group and dose levels.
To measure the Mood and Alertness of a marketed opioid analgesic versus placebo on alertness on quantitative pharmacodynamic experimental pain markers. | Change from Baseline (Pre-dose) in pressure pain thresholds and tolerance measurements at 46mins, 67 minutes
  Pressure pain threshold and tolerance measurements at 2 specified tender points reported by treatment group and dose levels. Mood and Alertness (Bond and Lader Visual Analogue Scale) presented graphically using box plots.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea